CLINICAL TRIAL: NCT06944366
Title: Comparing Exposure v Imagery Rescripting in People With Obsessive Compulsive Disorder (OCD): a Single Case Experimental Design (SCED)
Brief Title: Comparing Exposure v Imagery Rescripting in People With OCD: a SCED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRAS Project ID: 342003
Record Dates: First submitted 2025-04-03; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-01

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImR (Experimental): ImR completed as first intervention then ImExp
  Interventions: Other: Imagery intervention
- ImExp (Experimental): ImExp completed then ImR
  Interventions: Other: Imagery intervention

INTERVENTIONS:
Other: Imagery intervention — Imagery rescripting or imaginal exposure

SUMMARY:
Individuals with OCD may experience intrusive future orientated thoughts and images, which are extremely distressing and interfering in life. This project aims to explore whether imagery rescripting or exposure may be a more effective intervention for individuals with OCD experiencing such images.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* Main diagnosis of OCD (assessed by the Structured Clinical Interview for ICD11)
* Must report future orientated images that are distressing and ego-dystonic

Exclusion Criteria:

* Psychosis, bipolar disorder, or trauma disorder
* Current stimulant or hallucinogenic misuse, alcohol or substance misuse or dependence
* Intellectual disability, dementia, serious cognitive impairment, or organic brain disorder
* Personality Disorder as the main problem
* Active suicidality
* Concurrent engagement in other psychotherapy
* A patient may be taking anti-depressant medication so long as the dose has been stable for 6 weeks and there is no plan to increase the dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Obsessive Compulsive Inventory (OCI). | From the start of treatment until the end of treatment at 12 weeks.
  A 42-item self-report scale to assess the severity and type of OCD symptoms; the OCI uses a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely) and measures distress relating to 7 different subscales (washing, checking, doubting, ordering, obsessions, hoarding, and mental neutralizing). The total summed score of all items ranged between zero and 168. This measure will be completed at the beginning and end of each phase. Higher scores suggest more severe OCD symptomology.
Yale-Brown Obsessive-Compulsive scale (Y-BOCS). | From the start of treatment until the end of treatment at 12 weeks.
  A 10-item self-rated scale used to measure the severity of obsessive-compulsive symptoms and response to treatment; each item is scored from 0 (no symptoms) to 4 (extreme symptoms), with a total ranging from zero to 40. It will be completed at the beginning and end of each phase. Higher scores suggest more severe OCD symptomatology.
The Impact of Future Events Scale (IFES). | From the start of treatment until the end of treatment at 12 weeks.
  A 24-item self-rating scale used to measure the impact of intrusive prospective, personally relevant imagery. Each item is scored from 0 (no symptoms) to 4 (extreme symptoms), with a total ranging from zero to 96. Higher scores indicate greater symptomatology. This will be completed at the beginning and end of each phase.
The Florida Obsessive Compulsive Inventory (FOCI). | From the start of treatment until the end of treatment at 12 weeks.
  Designed to measure the severity and frequency of obsessive-compulsive symptoms in individuals. The severity scale (Part B) of the FOCI was used in the project. Part B is a 5-item self-rating scale used to measure the frequency, severity, and impact of obsessive-compulsive symptoms; each item is scored from 0 (no symptoms) to 4 (extreme symptoms), with a total ranging from zero to 20. Higher scores indicate greater symptomology.
Visual Analogue Scales (VAS). | From the start of treatment until the end of treatment at 12 weeks.
  Five daily self-report scales to be designed by the researchers using fixed scale (0=not at all; 10=extremely) answers to measure the following:
  Frequency of future orientated imagery Severity of future orientated imagery Vividness of future orientated imagery Degree of distress and aversive emotions associated with such imagery The urge to engage in compulsions/to neutralise the imagery.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Anxiety Disorders and Trauma, London, United Kingdom